CLINICAL TRIAL: NCT03959865
Title: Effectiveness and Persistence of Therapy With GLP-1 Receptor Agonists in Clinical Practice. A Multicenter Retrospective Study
Brief Title: GLP-1 REceptor Agonists and Real World EvIdeNce
Acronym: GLP-1REWIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Other Study IDs: 4462/AO/18
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Long-acting GLP-1RA: Patients who have been treated with weekly GLP-1RA (exenatide once weekly or dulaglutide)
  Interventions: Drug: Long-acting GLP-1RA
- Short-acting GLP-1RA: Patients who have been treated with daily GLP-1RA (exenatide bid or liraglutide or lixisenatide)
  Interventions: Drug: Short-acting GLP-1RA
- Human GLP-1 based GLP-1RA: Patients who have been treated with GLP-1RA based on human GLP-1 (dulaglutide or liraglutide)
  Interventions: Drug: Human-based GLP-1RA
- Exendin-based GLP-1RA: Patients who have been treated with weekly GLP-1RA (exenatide or lixisenatide)
  Interventions: Drug: Exendin-based GLP-1RA
- Fixed ratio combination of BI/GLP-1RA: Patients who have been treated with a fixed ratio combination of GLP-1RA and basal insulin (BI), such as IdegLira (insulin degludec / liraglutide) or IglarLixi (insulin glargine / lixisenatide)
  Interventions: Drug: Fixed ratio BI/GLP-1RA combination
- Flexible combination of BI/GLP-1RA: Patients who have been treated with any GLP-1RA in combination with any basal insulin (BI)
  Interventions: Drug: Flexible BI/GLP-1RA combination

INTERVENTIONS:
Drug: Long-acting GLP-1RA — Dulaglutide 0.75 or 1.5 mg /week or Exenatide once weekly 2 mg
  Groups: Long-acting GLP-1RA
Drug: Short-acting GLP-1RA — Liraglutide 0.6 mg or 1.2 mg or 1.8 mg / day or exenatide 10 mcg or 20 mcg bid or lixisenatide 10 mcg or 20 mcg / day.
  Groups: Short-acting GLP-1RA
Drug: Human-based GLP-1RA — Liraglutide 0.6 mg or 1.2 mg or 1.8 mg / day or dulaglutide 0.75 or 1.5 mg / week
  Groups: Human GLP-1 based GLP-1RA
Drug: Exendin-based GLP-1RA — Exenatide 10 mcg or 20 mcg day or 2 mg / week or lixisenatide 10 mcg or 20 mcg / day.
  Groups: Exendin-based GLP-1RA
Drug: Fixed ratio BI/GLP-1RA combination — Insulin degludec / liraglutide (0.036/U) or insulin glargine / lixisenatide (0.5 mcg/U)
  Groups: Fixed ratio combination of BI/GLP-1RA
Drug: Flexible BI/GLP-1RA combination — GLP-1RA (Liraglutide or dulaglutide or exenatide or lixisenatide) and basal insulin (BI, glargine, degludec, detemir, NPH insulin)
  Groups: Flexible combination of BI/GLP-1RA

SUMMARY:
Glucagon-like peptide-1 receptor agonists (GLP-1RA) are powerful second-line agents for the treatment of type 2 diabetes. GLP-1RA have bene marketed in 2010 in Italy and years of experience have accumulated for the treatment with this class of drugs. Cardiovascular outcome trials have shown that type 2 diabetic patients with established cardiovascular disease treated with GLP-1RA have a lower risk of future cardiovascular events.

In this real world study, we wish to evaluate retrospectively the effectiveness and persistence on treatment of GLP-1RA therapy in patients with type 2 diabetes from 2010 to 2018.

Effectiveness endpoints will be glycemic (fasting plasma glucose and HbA1c) and extra-glycemic (body weight and blood pressure). Data from diabetes outpatient clinics in North East Italy will be automatically extracted from electronic chart records and collected into a unique database.

Different groups of GLP-1RA therapies will be compared:

* Long-acting (e.g. dulaglutide and exenatide once weekly) versus short acting (exenatide, liraglutide and lixisenatide)
* Fixed versus flexible combinations of GLP-1RA and basal insulin.
* GLP-1RA with similarities to human GLP-1 (e.g. liraglutide) versus exendin-based GLP-1RA (e.g. exenatide).

DETAILED DESCRIPTION:
Introduction. Glucagon-like peptide-1 receptor agonists (GLP-1RA) are prioritized as a second-line therapy for the treatment of type 2 diabetes (T2D), especially in patients with a history of cardiovascular disease (CVD) or when there is a need to avoid weight gain and hypoglycemia. Randomized controlled trials (RCTs) have shown that addition of GLP-1RA is more effective in reducing HbA1c than addition of basal insulin (BI) in patients with uncontrolled T2D on oral therapy. GLP-1RA are associated with a low risk of hypoglycaemia and are provided with extra-glycemic effects, including reduction of body weight and blood pressure. Notably, GLP-1RA as a class improve cardiovascular outcomes in T2D patients with established CVD. These benefits justify the positioning of GLP-1RA as the first injectable therapy in most T2D patients and an alternative to insulin.

In the absence of data from RCTs, observational studies can provide medium-level evidence to inform clinical practice, if well-designed and carefully conducted. Real-world studies are hypothesis-generating and cannot substitute for RCTs, but they can guide the design of dedicated RCTs. Retrospective real-world studies are particularly attractive as they can rapidly gather data from large heterogeneous populations that are representative of those seen in routine clinical practice.

Design. The GLP-1REWIN study is a retrospective, multicenter, real-world study on T2D patients initiating GLP-1RA in the routine clinical practice of Italian diabetes outpatient clinics. The study will be conducted at 6 diabetes specialist outpatient clinics in the Veneto Region, North-East Italy.

Objective. The general objective of the study is to evaluate effectiveness of GLP-1RA on glycemic and extra-glycemic endpoints in the real world clinical practice from 2010 to 2018. The study will be conducted at diabetes Centers because only diabetologists were allowed to prescribe GLP-1RA in Italy during the study period.

Methods. Data will be collected retrospectively by automatically interrogating the same electronic chart at all Centers. A dedicated software was developed to extract all relevant anonymized patient information into a clinical research form without manual intervention. We will collect data on all patients aged 18-80 years, with a diagnosis of T2D since at least 1 year (as recorded in the chart), who initiated one GLP-1RA available on the market between 1st Jan 2010 to 31st Dec 2018. These included exenatide twice daily and once weekly, liraglutide, lixisenatide, dulaglutide and fixed ratio combinations of BI/GLP-1RA. The baseline visit date will be set as the date when the patients attended the outpatient clinic and received for the first time a new prescription of GLP-1RA. The following clinical characteristics and laboratory data will be collected from the electronic chart up to 90 days before baseline: age, sex, diabetes duration, body height and weight, body mass index (BMI), waist circumference, systolic and diastolic blood pressure (SBP and DBP), heart rate, fasting plasma glucose (FPG), HbA1c, total cholesterol, HDL cholesterol, triglycerides (LDL cholesterol was calculated using Friedwald's equation), liver enzymes, serum creatinine (eGFR was calculated using the chronic kidney diseae [CKD]-Epidemiology [EPI] equation), urinary albumin excretion rate (UAER, expressed as mg/g of urinary creatinine). Details on chronic complication, as reported by international classification of disease (ICD)-9 codes in the electronic charts wil be used to define the presence of micro- and macroangiopathy. Microangiopathy will be defined as any of the following: UAER >30 mg/g; eGFR<60 ml/min/1.73 m2; diabetic retinopathy (any stage) or diabetic macular edema; peripheral or autonomic neuropathy. Macroangiopathy will be defined as any of the following: peripheral arterial disease or peripheral revascularization; history of stroke/transient ischemic attack or carotid revascularization; ischemic heart disease, coronary artery disease, history of myocardial infarction, or coronary revascularization. Information on concomitant medications for the treatment of diabetes and of other cardiovascular risk factors will also be recorded. Detailed dose data will be collected for insulin and GLP-1RA. After having set the baseline date, we will identify the first available follow-up visit attended by the patients at the same Clinic at least 3 months after baseline. Updated values of HbA1c, FPG, SBP and body weight were recorded at the end of follow-up, along with updated information on medications and dosages of GLP-RA.

We will compare the changes in glycemic (HbA1c and fasting plasma glucose) and extra-glycemic (body weight and systolic blood pressure) effectiveness parameters between patients in two groups.

Different groups of GLP-1RA therapies will be compared:

* Long-acting (e.g. dulaglutide and exenatide once weekly) versus short acting (exenatide, liraglutide and lixisenatide)
* Fixed versus flexible combinations of GLP-1RA and basal insulin.
* GLP-1RA with similarities to human GLP-1 (e.g. liraglutide) versus exendin-based GLP-1RA (e.g. exenatide).

Statistics. Continuous variables will be expressed as mean ± standard deviation (SD) if normally distributed or as median (interquartile range) if non-normally distributed. Non-normal variables will be log-transformed before being analyzed with parametric tests. Categorical variables will be expressed as percentage. The comparison of baseline characteristics between two groups will be performed using unpaired 2-tail Student's t test for continuous variables and with chi square for categorical variables. To evaluate the balance between two groups, in addition to p-values, we will calculate the standardized mean difference (SMD). The intra-group change in effectiveness endpoint variables from baseline to end of follow-up will be analyzed using paired 2-tail Student's t test. We will then calculate the change in endpoint variables within each group, which will be compared using unpaired 2-tail Student's t test.

To address the issue of channeling bias (differences in baseline characteristics between the two groups that drive differential outcomes), we will use two different approaches. In the primary analysis, we will perform a propensity score matching (PSM), whereas multivariable adjustment (MVA) with linear regressions will be used as a second approach.

Statistical analyses will be performed using SAS version 9.4 (TS1M4) or higher and a 2-tail p-value <0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diabetes duration of at least 1 year
* Initiated on a GLP-1RA during the data collection period

Exclusion Criteria:

* Type 1 diabetes
* Previous therapy with a GLP-1RA before the data collection period

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients attending diabetes specialist clinics in North East Italy.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 3-12 months
  Change in HbA1c from baseline to end of follow-up

SECONDARY OUTCOMES:
Weight | 3-12 months
  Change in body weight from baseline to end of follow-up
Blood pressure | 3-12 months
  Change in systolic blood pressure from baseline to end of follow-up
Persistence | 3-12 months
  Percentage of patients who persist on treatment at the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Fadini, MD PhD, Study Chair — University of Padova
Locations (6):
- Italy (6):
  - Servizio di Diabetologia UOC Medicina Generale, Cittadella, Padova
  - U.O.S Diabetologia, Ospedale di Schiavonia, Monselice, Padova
  - U.O. Diabetologia ULSS2, Pieve di Soligo, Treviso
  - U.O. Diabetologia e Dietetica ULSS6, Padua
  - Azienda Ospedaliera di Padova, Padua
  - Diabetologia ULSS2, Treviso

IPD SHARING:
Plan to Share IPD: No
There is no possibility to share data with third parties.

REFERENCES:
- [Background] Lovshin JA, Drucker DJ. Incretin-based therapies for type 2 diabetes mellitus. Nat Rev Endocrinol. 2009 May;5(5):262-9. doi: 10.1038/nrendo.2009.48. PMID 19444259
- [Background] Bethel MA, Patel RA, Merrill P, Lokhnygina Y, Buse JB, Mentz RJ, Pagidipati NJ, Chan JC, Gustavson SM, Iqbal N, Maggioni AP, Ohman P, Poulter NR, Ramachandran A, Zinman B, Hernandez AF, Holman RR; EXSCEL Study Group. Cardiovascular outcomes with glucagon-like peptide-1 receptor agonists in patients with type 2 diabetes: a meta-analysis. Lancet Diabetes Endocrinol. 2018 Feb;6(2):105-113. doi: 10.1016/S2213-8587(17)30412-6. Epub 2017 Dec 6. PMID 29221659
- [Background] Davies MJ, D'Alessio DA, Fradkin J, Kernan WN, Mathieu C, Mingrone G, Rossing P, Tsapas A, Wexler DJ, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2018. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2018 Dec;41(12):2669-2701. doi: 10.2337/dci18-0033. Epub 2018 Oct 4. PMID 30291106
- [Background] Abd El Aziz MS, Kahle M, Meier JJ, Nauck MA. A meta-analysis comparing clinical effects of short- or long-acting GLP-1 receptor agonists versus insulin treatment from head-to-head studies in type 2 diabetic patients. Diabetes Obes Metab. 2017 Feb;19(2):216-227. doi: 10.1111/dom.12804. Epub 2016 Nov 29. PMID 27717195
- [Background] Singh S, Wright EE Jr, Kwan AY, Thompson JC, Syed IA, Korol EE, Waser NA, Yu MB, Juneja R. Glucagon-like peptide-1 receptor agonists compared with basal insulins for the treatment of type 2 diabetes mellitus: a systematic review and meta-analysis. Diabetes Obes Metab. 2017 Feb;19(2):228-238. doi: 10.1111/dom.12805. Epub 2016 Dec 5. PMID 27717130
- [Derived] Morieri ML, Rigato M, Frison V, Simioni N, D'Ambrosio M, Tadiotto F, Paccagnella A, Lapolla A, Avogaro A, Fadini GP. Fixed versus flexible combination of GLP-1 receptor agonists with basal insulin in type 2 diabetes: A retrospective multicentre comparative effectiveness study. Diabetes Obes Metab. 2019 Nov;21(11):2542-2552. doi: 10.1111/dom.13840. Epub 2019 Aug 12. PMID 31364233